CLINICAL TRIAL: NCT07029750
Title: Long-term Effects of Lipoabdominoplasty on Pulmonary Function and Sleep Apnea Risk in Obese Subjects
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Atlas University
Other Study IDs: auhucgun05
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Obstructive Sleep Apnea
Keywords: Obesity; Obstructive Sleep Apnea; Pulmonary Function; Lipoabdominoplasty
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive | interventions — Lipoabdominoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Obese subjects undergoing lipoabdominoplasty
  Interventions: Procedure: Lipoabdominoplasty

INTERVENTIONS:
Procedure: Lipoabdominoplasty — Combination of liposuction and abdominoplasty under general anesthesia. Klein solution used for tumescent liposuction. Muscle plication performed with 0 loop polydioxanone suture. Umbilicus preserved and repositioned. Postoperative compression corset used for 1 month.

SUMMARY:
This study investigates the long-term effects of lipoabdominoplasty on pulmonary function and obstructive sleep apnea (OSA) risk in obese patients. Participants were evaluated before and three months after surgery using spirometry, mMRC dyspnea scores, Epworth Sleepiness Scale (ESS), and STOP-Bang questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* BMI ≥ 30 kg/m²
* Eligible for lipoabdominoplasty
* Voluntary informed consent

Exclusion Criteria:

* Pregnancy
* Active pulmonary infections or chronic lung disease
* Additional surgical interventions during study period
* Refusal to participate or incomplete data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study will include adult patients (18-65 years) with a body mass index (BMI) over 30 kg/m² who are scheduled to undergo lipoabdominoplasty at a single tertiary care center. Eligible participants will be evaluated prior to surgery and again at 3 months postoperatively. Individuals with active pulmonary infections, chronic lung diseases, recent additional surgeries, or pregnancy will be excluded. All participants will provide written informed consent before enrollment. Approximately 24 participants are expected to complete both baseline and follow-up assessments.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 8-10 minutes
  Forced Vital Capacity will be measured before six-minute walk test according to the guideline of ERS.
Forced Expiratory Volume in 1 second (FEV1) | 8-10 minutes
  Forced Expiratory Volume in 1 second will be measured before six-minute walk test according to the guideline of ERS.
Peak Expiratory Flow (PEF) | 8-10 minutes
  Peak Expiratory Flow will be measured before six-minute walk test according to the guideline of ERS.
Forced Expiratory Flow 25-75% (FEF25-75) | 8-10 minutes
  Forced Expiratory Flow 25-75% will be measured before six-minute walk test according to the guideline of ERS.
mMRC Dyspnea Score | 8-10 minutes
  The dyspnea score will be assessed with the mMRC dyspnea score and is based on five stages of dyspnea caused by exertion and is scored between 0-4.
Sleep Apnea Risk Score | 8-10 minutes
  Sleep apnoea risk will be assessed using the Epworth Sleepiness Scale (ESS), a validated 8-item questionnaire that measures the subject's likelihood of falling asleep during daily activities. Higher scores reflect greater levels of daytime sleepiness and increased risk for conditions such as obstructive sleep apnoea.
Obstructive Sleep Apnea Risk Score | 8-10 minutes
  Obstructive sleep apnoea risk will be assessed assessed using the STOP-Bang questionnaire, an eight-item screening tool that evaluates snoring, tiredness, observed apnoea, high blood pressure, BMI, age, neck circumference, and gender. A higher score indicates a greater risk of OSA, with a cut-off of ≥3 commonly used to identify high-risk individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Hikmet Ucgun, PT, PhD, Principal Investigator — Atlas University
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No